CLINICAL TRIAL: NCT06556394
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability,Pharmacokinetics, and Pharmacodynamics of RAG-17 in Subjects With Amyotrophic Lateral Sclerosis (ALS) With Superoxide Dismutase Type 1 (SOD1) Gene Mutation
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RAG-17 in Subjects With Amyotrophic Lateral Sclerosis (ALS) With Superoxide Dismutase Type 1 (SOD1) Gene Mutation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ractigen Therapeutics. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RGN17-001
Record Dates: First submitted 2024-08-01; First posted 2024-08-16 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RAG-17 (Experimental): RAG-17 is administered by intrathecal injection to subjects with Amyotrophic Lateral Sclerosis (ALS) with Superoxide Dismutase Type 1 (SOD1) Gene Mutation
  Interventions: Drug: RAG-17
- Placebo (Placebo Comparator): Placebo is administered by intrathecal injection to subjects with Amyotrophic Lateral Sclerosis (ALS) with Superoxide Dismutase Type 1 (SOD1) Gene Mutation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RAG-17 — RAG-17 is a therapeutic small interfering RNA (siRNA).
  Arms: RAG-17
Drug: Placebo — Placebo will be administered via intrathecal injection
  Arms: Placebo

SUMMARY:
This is a Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RAG-17 in Subjects with Amyotrophic Lateral Sclerosis (ALS) with Superoxide Dismutase Type 1 (SOD1) Gene Mutation

DETAILED DESCRIPTION:
The study is a phase 1, randomized, double-blind, placebo controlled study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of RAG-17 in patients with Amyotrophic Lateral Sclerosis (ALS) with Superoxide Dismutase Type 1 (SOD1) gene mutation. The dose levels will be evaluated sequentially across separate cohorts using a rules-based design, wherein participants will receive RAG-17 or placebo at a ratio of 3:1.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily consents to participate in this study and provides written informed consent prior to the start of any study specific procedures.
2. ≥ 18 years of age at the time of informed consent.
3. Diagnosis of possible, laboratory supported probable, probable, or definite ALS according to the World Federation of Neurology El Escorial.
4. Documented SOD1 mutation.
5. Forced vital capacity (FVC) ≥50% of predicted value as adjusted for sex, age, and height (measured seated).
6. If taking riluzole or edaravone, subject must be on a stable dose or ≥30 days prior to Day 1 and expected to remain at that dose until the final study visit.

Exclusion Criteria:

1. Documented p.F21C SOD1 mutation.
2. Treatment with another investigational drug, biological agent, or device within 1 month or 5 half-lives of study agent, whichever is longer. Specifically, no prior treatment with small interfering ribonucleic acid, stem cell therapy, or gene therapy is allowed.
3. Current enrollment in any other interventional study.
4. History of or positive test result for human immunodeficiency virus, hepatitis C virus antibody or hepatitis B virus.
5. Pregnant or currently breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Adverse Events(AEs) | Before treatment and within 57 days after treatment
  Assesment of Safety and Tolerability: Incidence and severity of treatment-emergent Adverse Events(AEs) and Serious Adverse Events(SAEs)

SECONDARY OUTCOMES:
Plasma Pharmacokinetic (PK) Parameter: AUC0-last | Before treatment and within 48 hours after treatment
  Area Under the Plasma Concentration-Time Curve from Time 0 to the Last Measurable Non-zero Concentration
Plasma Pharmacokinetic (PK) Parameter: AUC0-inf | Before treatment and within 48 hours after treatment
  Area Under the Plasma Concentration-Time Curve from Time 0 Extrapolated to Infinity
Plasma Pharmacokinetic (PK) Parameter: Cmax | Before treatment and within 48 hours after treatment
  Peak Plasma Concentration
Plasma Pharmacokinetic (PK) Parameter: Tmax | Before treatment and within 48 hours after treatment
  Time to reach Cmax. If the maximum value occurs at more than one time point, Tmax is defined as the first time point with this value
Plasma Pharmacokinetic (PK) Parameter: λz | Before treatment and within 48 hours after treatment
  Elimination Rate Constant
Plasma Pharmacokinetic (PK) Parameter: T½ | Before treatment and within 48 hours after treatment
  Apparent Terminal Elimination Half-life of Study Drug
Plasma Pharmacokinetic (PK) Parameter: CL/F | Before treatment and within 48 hours after treatment
  Apparent Clearance
Plasma Pharmacokinetic (PK) Parameter: Vz/F | Before treatment and within 48 hours after treatment
  Apparent Volume of Distribution
Plasma Pharmacokinetic (PK) Parameter: MRT | Before treatment and within 48 hours after treatment
  Mean Residence Time
CSF Pharmacokinetic (PK) Parameter: Concentration | Before treatment and within 29 days after treatment
  Concentration in Cerebrospinal Fluid(CSF)
CSF Pharmacokinetic (PK) Parameter: T½ | Before treatment and within 29 days after treatment
  Half-life in Cerebrospinal Fluid(CSF)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Tiantan Hospital, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou